CLINICAL TRIAL: NCT01720199
Title: Diario Della Salute (DDS), a School-based Prevention Intervention to Promote Well-being for Grade 7 Students (12-13 Years)
Brief Title: A School-based Prevention Intervention to Promote Wellbeing in Preadolescents
Acronym: DDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale CN2 Alba-Bra (Other)
Collaborators: University of Eastern Piedmont (Other); Eclectica Sas di Beccaria Franca, Ermacora Antonella e C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCM2011-CUPJ19E11002100001
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Major Risk Factors for Noncommunicable Diseases
Keywords: universal prevention; primary prevention; health promotion; wellbeing; smoking; alcohol; diet; physical activity; emotional and social skills
MeSH Terms: conditions — Smoking; Motor Activity; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Preadolescents allocated to the Diario della Salute (DDS) intervention.
  Interventions: Other: Diario della Salute (DDS)
- Control group (No Intervention)

INTERVENTIONS:
Other: Diario della Salute (DDS) — DDS is composed by
  1. tools for children and their parents on health and social and emotional well-being issues:
     1. a diary for teens telling the story of four same-age students (e.g. experimenting with risky behaviors, conflicting feelings and thoughts, need for independence and control),
     2. a diary for parents telling the experience of a mum and a dad with teenage children (e.g. problems in the relationship with teenage children, family conflict, parental disappointment, etc.);
  2. five highly-standardized interactive lessons (2-4 hours each) on health issues administered by previously trained teachers.
  Arms: Intervention group

SUMMARY:
This is a field study aiming to evaluate a school-based prevention intervention, Diario della Salute (DDS).

DETAILED DESCRIPTION:
Diario della Salute (DDS) is a school-based prevention intervention based on the following theories:

1. social-cognitive theory (Bandura, 1977; 1986)
2. theory of multiple intelligences (Gardner, 1987)
3. emotional intelligence theory (Goleman, 1997)
4. theory of planned behavior (Ajzen, 1991)
5. transtheoretical model of change (Prochaska, Diclemente, 1982; 1992).

DDS is composed by:

1. tools for children and their parents on health and social and emotional well-being issues:

   1. a diary for teens telling the story of four same-age students (e.g. experimenting with risky behaviors, conflicting feelings and thoughts, need for independence and control),
   2. a diary for parents telling the experience of a mum and a dad with teenage children (e.g. problems in the relationship with teenage children, family conflict, parental disappointment, etc.);
2. five highly-standardized interactive lessons (2-4 hours each) on health issues administered by previously trained teachers.

Assignment of schools to study arms (DDS intervention vs. no intervention) will be cluster-randomized. Schools will be matched by number of students and average socioeconomic status. In some study areas schools will not be allocated by chance, but they will be analyzed separately from other schools.

Two anonymous surveys focusing on main outcomes (wellbeing, tobacco smoking, alcohol, physical activity and diet) will be before and after the intervention. Pre and post surveys will be linked through an anonymous code (Galanti, 2006).

ELIGIBILITY:
Inclusion Criteria:

* schools providing consensus to study participation

Exclusion Criteria:

* schools involved in structured prevention programs with similar objectives

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2630 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Self-reported Social And Emotional Well-Being | Past 30 Days
  Subjective well-being is defined as 'a person's cognitive and affective evaluations of his or her life' (Diener, Lucas, & Oshi, 2002, p. 63).

SECONDARY OUTCOMES:
Self-reported Cigarette Use | Past 30 Days
  Frequency of cigarette smoking
Self-reported Drunkenness Episode(s) | Past 30 Days
  Frequency of drunkenness episodes
Self-reported Dietary Habits | Past 30 Days
  Consumption of beverages and foods such as pop drinks, chips, vegetables, fruits and others
Self-reported Frequency of Physical Exercise | Past 30 Days
  Frequency of moderate and heavy physical exercise
Self-reported Physical and Verbal Aggression | Past 30 Days
  Aggression is generally defined as behaviors that are intended to hurt or harm others by damaging their physical and psychological well-being and includes physically and verbally aggressive behaviors such as hitting, pushing, kicking, and threatening, etc (Dodge et al. 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Faggiano, MD, Principal Investigator — University of Eastern Piedmont; Antonella Ermacora, MSc, Study Chair — Eclectica Sas di Beccaria Franca, Ermacora Antonella e C.; Elias Allara, MD, Study Director — University of Eastern Piedmont
Locations (1):
- Azienda Sanitaria Locale CN2 Alba-Bra, Alba, Cuneo, Italy

REFERENCES:
- [Background] Ajzen, I. (1991). The theory of planned behavior. Organizational Behavior and Human Decision Processes, 50, 179-211.
- [Background] Bandura, A. (1977). Social Learning Theory. New York: General Learning Press.
- [Background] Bandura, A. (1986). Social Foundations of Thought and Action. Englewood Cliffs, NJ: Prentice-Hall.
- [Background] Dodge, K.A., Coie, J.D., & Lynam, D. (2006). Aggression and antisocial behavior in youth. In W. Damon (Series Ed.), & N. Eisenberg (Vol. Ed.) (Ed.). Handbook of Child Psychology, Vol. 3: Social, Emotional, and Personality Development6th edition (pp. 719-788). Wiley.
- [Background] Galanti MR, Siliquini R, Cuomo L, Melero JC, Panella M, Faggiano F; EU-DAP study group. Testing anonymous link procedures for follow-up of adolescents in a school-based trial: the EU-DAP pilot study. Prev Med. 2007 Feb;44(2):174-7. doi: 10.1016/j.ypmed.2006.07.019. Epub 2006 Sep 18. PMID 16979751
- [Background] Gardner, H. (1987). Beyond a modular view of mind. In W. Damon (Ed.), New Directions for Child Development, Tenth Anniversary Edition. Also in W. Damon (Ed.) (1988), Child Development Today and Tomorrow (222-239). San Francisco: Jossey-Bass.
- [Background] Goleman, D. (1998). Working with emotional intelligence. New York: Bantam.
- [Background] Prochaska J.O. and DiClemente C.C. (1982). Trans-theoretical therapy - toward a more integrative model of change. Psychotherapy: Theory, Research and Practice 19(3):276-288
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- See also: Project website (in Italian). — http://www.diariodellasalute.it/